CLINICAL TRIAL: NCT00501059
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Parallel Group Study to Assess the Efficacy (Reduction of Cardiovascular Disease Events) and Safety of 100 mg Enteric-Coated Acetylsalicylic Acid in Patients at Moderate Risk of Cardiovascular Disease
Brief Title: A Study to Assess the Efficacy and Safety of Enteric-Coated Acetylsalicylic Acid in Patients at Moderate Risk of Cardiovascular Disease
Acronym: ARRIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12198; 2006-003622-29 (EudraCT Number)
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-09

CONDITIONS: Moderate Risk of CVD
Keywords: Primary prevention of coronary heart disease; Stroke and cardiovascular death; Aspirin
MeSH Terms: conditions — Stroke | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetylsalicylic acid (Aspirin, BAYE4465) (Experimental): Participants received 1 tablet of enteric-coated acetylsalicylic acid [100 milligram (mg)] orally once daily.
  Interventions: Drug: Aspirin (Acetylsalicylic acid, BAYE4465)
- Placebo (Placebo Comparator): Participants received 1 tablets of matching placebo orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin (Acetylsalicylic acid, BAYE4465) — 100mg enteric coated Aspirin, taken daily
  Arms: Acetylsalicylic acid (Aspirin, BAYE4465)
Drug: Placebo — Placebo, taken daily
  Arms: Placebo

SUMMARY:
The use of acetylsalicylic acid in the primary prevention of cardiovascular events has been extensively studied but to a lesser extent in patients with moderate levels of cardiovascular risk. The current study is designed to prove the efficacy and tolerability of 100 mg enteric-coated Aspirin versus placebo in the prevention of cardiovascular disease (CVD) events, which include fatal and nonfatal myocardial infarction, fatal and nonfatal stroke and CV death, in a population with no history of known CVD who are at moderate risk of major CHD events (approximately 10-20% 10 year CHD risk). This corresponds to a patient population mean 10-year CVD risk of approximately 30%. Subjects are treated in a standard care setting and may receive treatment for the underlying risk factors as defined by the treating physician. Outcome events will be adjudicated by an Endpoint Adjudication Committee and the study will be monitored by an independent Data Safety Monitoring Board.

DETAILED DESCRIPTION:
Summary of substantial Protocol amendments

Amendment #2 from 09-APR-2008:

* Systolic blood pressure (SBP) limit of 170 mmHg has been added to the exclusion criteria
* Exclusion of patients currently taking anticoagulant medication
* A longer interval between the daily dose of study drug and ibuprofen
* Revised wording in moderate risk definitions for coronary heart disease (CHD) and cerebrovascular disease (CVD): "To evaluate the clinical effects of a 100 mg/day enteric-coated acetylsalicylic acid versus placebo in the reduction of CVD events in patients at moderate risk of major CHD events (approximately 10 to 20% 10-year CHD risk; approximately 20 to 30% 10-year risk of CVD). This corresponds to a patient population mean 10-year CVD risk of approximately 30%."

Amendment #3 from 02-JAN-2009

• Increase in the number of allowed risk factors for males, age is no longer a risk factor

Amendment #4 from 02-OCT-2013

* The primary endpoint is changed to include confirmed UA and TIA.
* The estimated event rate is changed to 1.5% per year due to new information.
* Effect size (risk reduction) changed from 14.9% to 17 to 18%.
* Achieving 60,000 person-years instead of 1488 primary endpoint events
* Additional treatment and follow-up for a maximum of another 12 months.
* Change to reduced adverse event and concomitant therapy reporting

ELIGIBILITY:
Inclusion Criteria:

* Males aged 55 years and above with 2 to 4 risk factors. Male Risk Factors:

  * Elevated cholesterol (Tchol>200 mg/dL or LDL>130 mg/dL; as measured at screening) irrespective of current treatment
  * Current smoking: defined as any cigarette smoking in the past 12 months
  * Low HDL cholesterol (HDL<40 mg/dL; as measured at screening)
  * Elevated blood pressure (SBP>140 mmHg; as measured at screening)
  * Currently on any medication to treat high blood pressure
  * Positive family history of early CHD (a first-degree relative [father, mother, brother, sister, son, daughter] suffered a heart attack [myocardial infarction] before the age of 60 years)
* Females aged 60 and above with 3 or more risk factors. Female Risk Factors:

  * Elevated cholesterol (Tchol>240 mg/dL or LDL>160 mg/dL; as measured at screening) irrespective of current treatment
  * Current smoking: defined as any cigarette smoking in the past 12 months
  * Low HDL cholesterol (HDL<40 mg/dL; as measured at screening)
  * Elevated blood pressure (SBP>140 mmHg; as measured at screening)
  * Currently on any medication to treat high blood pressure
  * Positive family history of early CHD (a first-degree relative [father, mother, brother, sister, son, daughter] suffered a heart attack [myocardial infarction] before the age of 60 years)
* An understanding and willingness to comply with trial procedures and has given written informed consent to participate in the trial

Exclusion Criteria:

* History of a documented vascular event, such as MI, stroke, coronary artery angioplasty or stenting, coronary artery bypass graft, relevant arrhythmias, or congestive heart failure or vascular intervention
* Patients who are at higher than moderate risk on the basis of their diabetes status, other factors known to the investigator, or the currently used national risk score
* Known contraindications to the study drug, e.g. hypersensitivity to acetylsalicylic acid
* Recent (in the past year) history of gastrointestinal or genitourinary bleeding or other bleeding disorders
* Active diagnosed and documented reflux esophagitis
* Patients presenting with any medical condition, or psychiatric or substance abuse disorder, that, in the opinion of the investigator, is likely to affect the patient's ability to complete the study or precludes the patient's participation in the study
* Lactating women or women of childbearing potential
* Severe liver disease or damage based on the clinical judgment of the investigator
* Severe renal disease or damage based on the clinical judgement of the investigator
* A definite indication for acetylsalicylic acid therapy, other antiplatelet drug, or anticoagulant in the opinion of the physician
* A history of asthma induced by administration of salicylates or substances with a similar action, notably NSAIDS
* Chronic, frequent (> 5 days/month) use of NSAIDs (including aspirin, or aspirin containing products), COX-2 inhibitors or metamizole
* Current participation in any other trials involving investigational products within 30 days prior to the Screening Visit
* Current use of an anticoagulant medication
* Sitting systolic blood pressure greater than 170 mmHg

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12546 (Actual)
Dates: Start 2007-07-05 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (380):
- United States (71):
  - Birmingham, Alabama
  - Graysville, Alabama
  - Pell City, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Fremont, California
  - Huntington Park, California
  - Los Angeles, California
  - Rancho Cucamonga, California
  - Rolling Hills Estates, California
  - Helping Hands Clinical Trials, Santa Ana, California
  - Newark, Delaware
  - Medical Research Trust, Boynton Beach, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Medical Research Centers of South Florida, Inc., Hollywood, Florida
  - Office of Dr.Larry Levinson, DO, Hollywood, Florida
  - Kissimmee, Florida
  - Largo, Florida
  - Marianna, Florida
  - Panama City, Florida
  - Tallahassee Memorial Family, Quincy, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Lockport, Illinois
  - Vernon Hills, Illinois
  - Evansville, Indiana
  - Fort Wayne, Indiana
  - Lebanon, Kentucky
  - Prince Frederick, Maryland
  - Bridgman, Michigan
  - Cadillac, Michigan
  - Interlochen, Michigan
  - Troy, Michigan
  - Port Gibson, Mississippi
  - Florissant, Missouri
  - Broken Bow, Nebraska
  - Omaha, Nebraska
  - Belvidere, New Jersey
  - Cherry Hill, New Jersey
  - Clifton, New Jersey
  - Hainesport, New Jersey
  - Jersey City, New Jersey
  - Lawrenceville, New Jersey
  - Linden, New Jersey
  - PharmaTrials, Inc., Perth Amboy, New Jersey
  - Stratford, New Jersey
  - Burlington, North Carolina
  - Columbus, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Carlisle, Ohio
  - Marion, Ohio
  - Montgomery, Ohio
  - Perrysburg, Ohio
  - Doylestown, Pennsylvania
  - Duncansville, Pennsylvania
  - Sellersville, Pennsylvania
  - Taylors, South Carolina
  - Daingerfield, Texas
  - McKinney, Texas
  - Rockwall, Texas
  - San Antonio, Texas
  - San Marcos, Texas
  - Stephenville, Texas
  - Sugar Land, Texas
  - Honaker, Virginia
  - Merit Medical Group, Inc., Richlands, Virginia
- Germany (112):
  - Benningen am Neckar, Baden-Wurttemberg
  - Deggingen, Baden-Wurttemberg
  - Dossenheim, Baden-Wurttemberg
  - Ettlingen, Baden-Wurttemberg
  - Graben-Neudorf, Baden-Wurttemberg
  - Heilbronn, Baden-Wurttemberg
  - Hockenheim, Baden-Wurttemberg
  - Ludwigsburg, Baden-Wurttemberg
  - Schwetzingen, Baden-Wurttemberg
  - Sinzheim, Baden-Wurttemberg
  - Stockach, Baden-Wurttemberg
  - Stuttgart, Baden-Wurttemberg
  - Trossingen, Baden-Wurttemberg
  - Weinheim, Baden-Wurttemberg
  - Arzberg, Bavaria
  - Bergrheinfeld, Bavaria
  - Dinkelsbühl, Bavaria
  - Gars, Bavaria
  - Hohenau, Bavaria
  - Künzing, Bavaria
  - München, Bavaria
  - Oberaurach, Bavaria
  - Sand Am Main, Bavaria
  - Schrobenhausen, Bavaria
  - Spalt, Bavaria
  - Straßkirchen, Bavaria
  - Sulzbach-Rosenberg, Bavaria
  - Ursensollen, Bavaria
  - Cottbus, Brandenburg
  - Elsterwerda, Brandenburg
  - Gransee, Brandenburg
  - Ketzin, Brandenburg
  - Potsdam, Brandenburg
  - Frankfurt am Main, Hesse
  - Hanau, Hesse
  - Kelkheim, Hesse
  - Rotenburg an der Fulda, Hesse
  - Wetter, Hesse
  - Aurich, Lower Saxony
  - Bockenem, Lower Saxony
  - Braunschweig, Lower Saxony
  - Horneburg, Lower Saxony
  - Jühnde, Lower Saxony
  - Loxstedt, Lower Saxony
  - Nienburg, Lower Saxony
  - Northeim, Lower Saxony
  - Papenburg, Lower Saxony
  - Stuhr, Lower Saxony
  - Wardenburg, Lower Saxony
  - Weyhe, Lower Saxony
  - Winsen, Lower Saxony
  - Aachen, North Rhine-Westphalia
  - Arnsberg, North Rhine-Westphalia
  - Bad Lippspringe, North Rhine-Westphalia
  - Bad Salzuflen, North Rhine-Westphalia
  - Bad Sassendorf, North Rhine-Westphalia
  - Bergkamen, North Rhine-Westphalia
  - Bochum, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Dortmund, North Rhine-Westphalia
  - Duisburg, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Freudenberg, North Rhine-Westphalia
  - Greven, North Rhine-Westphalia
  - Hamm, North Rhine-Westphalia
  - Hünxe, North Rhine-Westphalia
  - Kamp-Lintfort, North Rhine-Westphalia
  - Krefeld, North Rhine-Westphalia
  - Langenfeld, North Rhine-Westphalia
  - Lienen, North Rhine-Westphalia
  - Lippetal, North Rhine-Westphalia
  - Löhne, North Rhine-Westphalia
  - Marl, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Netphen, North Rhine-Westphalia
  - Porta Westfalica, North Rhine-Westphalia
  - Remscheid, North Rhine-Westphalia
  - Siegen, North Rhine-Westphalia
  - Viersen, North Rhine-Westphalia
  - Welver, North Rhine-Westphalia
  - Wetter, North Rhine-Westphalia
  - Witten, North Rhine-Westphalia
  - Kallstadt, Rhineland-Palatinate
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Nassau, Rhineland-Palatinate
  - Rhaunen, Rhineland-Palatinate
  - Speyer, Rhineland-Palatinate
  - Beucha, Saxony
  - Borna, Saxony
  - Delitzsch, Saxony
  - Dresden, Saxony
  - Leipzig, Saxony
  - Markkleeberg, Saxony
  - Meissen, Saxony
  - Oberwiesenthal, Saxony
  - Riesa, Saxony
  - Wermsdorf, Saxony
  - Bitterfeld-Wolfen, Saxony-Anhalt
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Bad Bramstedt, Schleswig-Holstein
  - Reinfeld, Schleswig-Holstein
  - Apolda, Thuringia
  - Blankenhain, Thuringia
  - Grimma, Thuringia
  - Berlin
  - Daaden
  - Hamburg
  - Rehburg-Loccum
  - Riede
  - Thedinghausen
- Ireland (9):
  - Bishopstown, Cork
  - Kilmallock, Limerick
  - Rathkeale, Limerick
  - Tallow, Waterford
  - Enniscorthy, Wexford
  - Gorey, Wexford
  - Bray, Wicklow
  - Cork
  - Dublin
- Italy (19):
  - Chieti, Abruzzo
  - Foggia, Apulia
  - Amandola, Ascoli Piceno
  - Napoli, Campania
  - Reggio Emilia, Emilia-Romagna
  - Chiavari, Genova
  - Rome, Lazio
  - Como, Lombardy
  - Varese, Lombardy
  - Legnano, Milano
  - Novara, Piedmont
  - Turin, Piedmont
  - Catania, Sicily
  - Chieri, Torino
  - Moncalieri, Torino
  - Grosseto, Tuscany
  - Asti
  - Bergamo
  - Reggio Emilia
- Poland (35):
  - Bialystok
  - Bydgoszcz
  - Chrzanów
  - Czechowice-Dziedzice
  - Elblag
  - Gdansk
  - Gdynia
  - Gliwice
  - Grodzisk Mazowiecki
  - Katowice
  - Krakow
  - Kutno
  - Linia
  - Lodz
  - Lublin
  - Malbork
  - Małaszewicze
  - Nakło nad Notecią
  - Olkusz
  - Ostrów Wielkopolski
  - Poznan
  - Przeworsk
  - Radom
  - Skierniewice
  - Sobótka
  - Sopot
  - Szczyrk
  - Warsaw
  - Wąbrzeźno
  - Wejherowo
  - Wola
  - Wroclaw
  - Włocławek
  - Zabrze
  - Łańcut
- Puerto Rico (5):
  - Guaynabo
  - Manatí
  - Orocovis
  - San Juan
  - Trujilo Alto
- Spain (28):
  - Sobrado Dos Monxes, A Coruña
  - La Roda, Albacete
  - Benidorm, Alicante
  - Elche, Alicante
  - Petrel, Alicante
  - Xixona, Alicante
  - Vic (Barcelona), Catalonia
  - Begonte, Lugo
  - Viveiro, Lugo
  - Espinardo, Murcia
  - Ourense, Ourense
  - Oviedo, Principality of Asturias
  - Posada de Llanes, Principality of Asturias
  - Gümar, Santa Cruz De Tenerife
  - La Victoria, Santa Cruz De Tenerife
  - Alcover, Tarragona
  - Albacete
  - Alicante
  - Badajoz
  - Barcelona
  - Huelva
  - León
  - Lugo
  - Madrid
  - Murcia
  - Salamanca
  - Santander
  - Valladolid
- United Kingdom (101):
  - Ballymena, Antrim
  - Crumlin, Antrim
  - Newtonabbey, Antrim
  - Craigavon, Armagh
  - Bath, Avon
  - Radstock, Avon
  - Irvine, Ayrshire
  - Luton, Bedfordshire
  - Slough, Berkshire
  - Ely, Cambridgeshire
  - Peterborough, Cambridgeshire
  - Sandbach, Cheshire
  - Boscastle, Cornwall
  - Fowey, Cornwall
  - Penzance, Cornwall
  - Saltash, Cornwall
  - St Austell, Cornwall
  - Chesterfield, Derbyshire
  - Dronfield, Derbyshire
  - Plymouth, Devon
  - Carryduff, Down
  - Annan, Dumfries And Galloway
  - Bishop Auckland, Durham
  - Darlington, Durham
  - Leigh-on-Sea, Essex
  - Tiptree, Essex
  - High Valleyfield, Fife
  - Glasgow, Glasgow City
  - Bangor, Gwynedd
  - Hitchin, Hertfordshire
  - Letchworth Garden City, Hertfordshire
  - Canterbury, Kent
  - Chestfield, Kent
  - Whitstable, Kent
  - Carstairs, Lanarkshire
  - Coatbridge, Lanarkshire
  - Forth, Lanarkshire
  - Blackpool, Lancashire
  - Bolton, Lancashire
  - Hinckley, Leicestershire
  - Wells-next-the-Sea, Norfolk
  - Wymondham, Norfolk
  - Antrim, North Ireland
  - Tyrone, North Ireland
  - Wellingborough, Northamptonshire
  - Chipping Norton, Oxfordshire
  - Eccles, Sheffield
  - Bath, Somerset
  - Barry, SOuth Glamorgan
  - Doncaster, South Yorkshire
  - Sheffield, South Yorkshire
  - Chapelhall, Stratchclyde
  - Glasgow, Stratchclyde
  - Hamilton, Stratchclyde
  - Johnstone, Stratchclyde
  - Motherwell, Stratchclyde
  - Bury Saint Edmonds, Suffolk
  - Bury St Edmunds, Suffolk
  - Hadleigh, Suffolk
  - Stowmarket, Suffolk
  - Addlestone, Surrey
  - East Horsley, Surrey
  - Worcester Park, Surrey
  - Newcastle upon Tyne, Tyne and Wear
  - Coventry, Warwickshire
  - Rugby, Warwickshire
  - Coventry, West Midlands
  - Brighton, West Sussex
  - Crawley, West Sussex
  - Leeds, West Yorkshire
  - Bradford-on-Avon, Wiltshire
  - Chippenham, Wiltshire
  - Corsham, Wiltshire
  - Trowbridge, Wiltshire
  - Westbury, Wiltshire
  - Aberdeen
  - Airedire
  - Antrim
  - Bath
  - Belfast
  - Bellshill
  - Blantyre
  - Cardiff
  - Coatrbridge
  - Crossgar
  - Doncaster
  - Dundee
  - Glasgow
  - Hamilton
  - Inverness
  - Ipswich
  - Lockerbie
  - London
  - Manchester
  - New Stevenson
  - Paisley
  - Peterborough
  - Thornhill
  - Watford
  - Wishaw
  - Witley Bay

REFERENCES:
- [Result] Gaziano JM, Brotons C, Coppolecchia R, Cricelli C, Darius H, Gorelick PB, Howard G, Pearson TA, Rothwell PM, Ruilope LM, Tendera M, Tognoni G; ARRIVE Executive Committee. Use of aspirin to reduce risk of initial vascular events in patients at moderate risk of cardiovascular disease (ARRIVE): a randomised, double-blind, placebo-controlled trial. Lancet. 2018 Sep 22;392(10152):1036-1046. doi: 10.1016/S0140-6736(18)31924-X. Epub 2018 Aug 26. PMID 30158069
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 15823 subjects were screened. Of these, 3277 subjects were screening failures. The remaining 12546 subjects were randomized to treatment.
Groups:
- Acetylsalicylic Acid (Aspirin, BAYE4465): Subjects received 1 tablet of enteric-coated acetylsalicylic acid [100 milligram (mg)] orally once daily.
- Placebo: Subjects received 1 tablets of matching placebo orally once daily.
Period: Overall Study
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) | Placebo
Started | 6270 | 6276
Completed | 4402 | 4384
Not Completed | 1868 | 1892
Not completed — Protocol Violation | 80 | 69
Not completed — Death | 140 | 137
Not completed — Other | 236 | 239
Not completed — Missing end-of-study page | 91 | 92
Not completed — Clinical endpoint reached | 110 | 123
Not completed — Insufficient therapeutic effect | 4 | 5
Not completed — Consent withdrawn by subject | 817 | 873
Not completed — Non-compliant with study treatment | 23 | 16
Not completed — Reason not given | 3 | 1
Not completed — Adverse Event | 129 | 122
Not completed — Lost to Follow-up | 210 | 198
Not completed — Not treated | 25 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) | Placebo | Total
Number analyzed (Participants) | 6270 | 6276 | 12546
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (7.10) | 63.9 (7.05) | 63.9 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1851 | 1857 | 3708
  Male | 4419 | 4419 | 8838

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Occurrence of the Composite Outcome of MI (Myocardial Infarction), Stroke, Cardiovascular Death, UA (Unstable Angina) or TIA (Transient Ischemic Attack)
Description: The primary efficacy endpoint was a composite outcome consisting of the first occurrence of confirmed MI, stroke, cardiovascular death, UA, TIA. The time to event was defined as the number of days from the date of randomization to the date of the event confirmed by adjudication. The numbers of days for milestones when 1%, 2%, 3% and 4% of the subjects have reached endpoint events were estimated from Kaplan-Meier-Analyses.
Time Frame: Until follow-up (approximate 6 years)
Population: Intention-to-treat. The intent-to-treat (ITT) group (N=12546) consists of all patients who were randomized to the assigned study drug.
Measure: Count of Units; unit: Days
Units Other Than Participants: Days
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) | Placebo
Number analyzed (Participants) | 6270 | 6276
Number analyzed (Days) | 1630 | 1630
Days
  Days until 1% subjects had an efficacy event | 528 | 381
  Days until 2% subjects had an efficacy event | 889 | 796
  Days until 3% subjects had an efficacy event | 1225 | 1134
  Days until 4% subjects had an efficacy event | 1630 | 1582
Statistical Analysis 1: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Primary efficacy analysis of time to the composite endpoint was conducted via a 2-sided log-rank test stratified for treatment, country, and sex. Results would be considered statistically significant and the primary objective of the study will have been met if the 2-sided P value is ≤0.05; Test type: Superiority or Other; p = 0.597, Log Rank

2. Secondary Outcome: Time to the First Occurrence of the Composite Outcome of Cardiovascular Death, MI, or Stroke (Ischemic, Hemorrhagic, or Unknown)
Description: The time to Composite outcome consisting of the first occurrence of cardiovascular death, MI, or stroke (ischemic, hemorrhagic, or unknown) was defined as the number of days from the date of randomization to the date of the event confirmed by adjudication. The numbers of days for milestones when 1%, 2%, 3% and 4% of the subjects have reached endpoint events were estimated from Kaplan-Meier-Analyses.
Time Frame: Until follow-up (approximate 6 years)
Population: ITT
Measure: Count of Units; unit: Days
Units Other Than Participants: Days
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) | Placebo
Number analyzed (Participants) | 6270 | 6276
Number analyzed (Days) | 1949 | 1949
Days
  Days until 1% subjects had an efficacy event | 678 | 522
  Days until 2% subjects had an efficacy event | 1167 | 1053
  Days until 3% subjects had an efficacy event | 1599 | 1501
  Days until 4% subjects had an efficacy event | 1949 | 1930
Statistical Analysis 1: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Statistics for time to the composite endpoint was conducted via a 2-sided log-rank test stratified for treatment, country, and sex. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Superiority or Other; p = 0.6125, Log Rank

3. Secondary Outcome: Time to the First Occurrence of the Individual Components of the Primary: Non-fatal MI, Total MI, Non-fatal Stroke, Total Stroke, Cardiovascular Death, UA and TIA
Description: The time to event was defined as the number of days from the date of randomization to the date of the event confirmed by adjudication. The numbers of days for milestones when 1%, 2%, 3% and 4% of the subjects have reached endpoint events were estimated from Kaplan-Meier-Analyses.
Time Frame: Until follow-up (approximately 6 years)
Population: ITT
Measure: Count of Units; unit: Days
Units Other Than Participants: Days
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) | Placebo
Number analyzed (Participants) | 6270 | 6276
Number analyzed (Days) | 2128 | 2128
Days
  Days until 1% subjects had non-fatal MI | 1309 | 1085
  Days until 2% subjects had non-fatal MI | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | 2121
  Days until 1% subjects had total MI | 1216 | 1014
  Days until 2% subjects had total MI | 2128 | 1906
  Days until 1% subjects had non-fatal stroke | 1576 | 1650
  Days until 2% subjects had non-fatal stroke | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study.
  Days until 1% subjects had total stroke | 1543 | 1627
  Days until 2% subjects had total stroke | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study.
  Days until 1% subjects had cardiovascular death | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study.
  Days until 2% subjects had cardiovascular death | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study.
  Days until 1% subjects had UA | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study.
  Days until 2% subjects had UA | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study.
  Days until 1% subjects had TIA | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study.
  Days until 2% subjects had TIA | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study..
Statistical Analysis 1: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Statistics for time to non-fatal MI was conducted via a 2-sided log-rank test stratified for treatment, country, and sex. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Superiority or Other; p = 0.4505, Log Rank
Statistical Analysis 2: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Statistics for time to total MI was conducted via a 2-sided log-rank test stratified for treatment, country, and sex. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Superiority or Other; p = 0.229, Log Rank
Statistical Analysis 3: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Statistics for time to total non-fatal stroke was conducted via a 2-sided log-rank test stratified for treatment, country, and sex. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Superiority or Other; p = 0.3947, Log Rank
Statistical Analysis 4: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Statistics for time to total stroke was conducted via a 2-sided log-rank test stratified for treatment, country, and sex. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Superiority or Other; p = 0.5125, Log Rank

4. Secondary Outcome: Time to All-cause Mortality, the First Occurrence of All Cancers Excluding Non-melanoma Skin Cancer (NMSC) and the First Occurrence of Colon Cancer
Description: as for outcome 3
Time Frame: Until follow-up (approximately 6 years)
Population: ITT
Measure: Count of Units; unit: Days
Units Other Than Participants: Days
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) | Placebo
Number analyzed (Participants) | 6270 | 6276
Number analyzed (Days) | 1970 | 1970
Days
  Days until 1% subjects had all-cause mortality | 838 | 938
  Days until 2% subjects had all-cause mortality | 1493 | 1460
  Days until 3% subjects had all-cause mortality | 1970 | 1963
  Days until 4% subjects had all-cause mortality | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study.
  Days until 1% subjects had all cancer excl. NMSC | 374 | 420
  Days until 2% subjects had all cancer excl. NMSC | 849 | 805
  Days until 3% subjects had all cancer excl. NMSC | 1164 | 1276
  Days until 4% subjects had all cancer excl. NMSC | 1542 | 1751
  Days until 1% subjects had colon cancer | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study.
  Days until 2% subjects had colon cancer | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study..
  Days until 3% subjects had colon cancer | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study.
  Days until 4% subjects had colon cancer | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study. | NA — Not applicable (NA) indicates that these milestones did not occur before completion of the study..
Statistical Analysis 1: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of time to all-cause mortality was conducted via a 2-sided log-rank test stratified for treatment, country, and sex. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Superiority or Other; p = 0.9544, Log Rank
Statistical Analysis 2: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of time to the first occurrence of all cancers excluding non-melanoma skin cancer was conducted via a 2-sided log-rank test stratified for treatment, country, and sex. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Superiority or Other; p = 0.4422, Log Rank
Statistical Analysis 3: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of time to the first occurence colon cancer was conducted via a 2-sided log-rank test stratified for treatment, country, and sex. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Superiority or Other; p = 0.611, Log Rank

5. Secondary Outcome: Incidence of All-cause Mortality, All Cancers Excluding Non-melanoma Skin Cancer and Colon Cancer
Time Frame: Until follow-up (approximately 6 years)
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) | Placebo
Number analyzed (Participants) | 6270 | 6276
Percentage of participants
  all-cause mortality | 2.55 | 2.57
  all cancers excluding non-melanoma skin cancer | 4.02 | 3.76
  colon cancer | 0.48 | 0.41
Statistical Analysis 1: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of incidence of all-cause mortality was conducted via a 2-sided log-rank test. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Other; p = 0.9459, Log Rank; Cox Proportional Hazard = 0.99, 95% CI 2-sided [0.80 to 1.24]

6. Secondary Outcome: Incidence of Confirmed MI, Stroke, Cardiovascular Death, UA, and TIA Separately
Description: The percentages of subjects with the efficacy endpoints of confirmed MI, stroke, cardiovascular death, UA and TIA are reported separately. *all other CV death without fatal MI and fatal stroke
Time Frame: Until follow-up (approximately 6 years)
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) | Placebo
Number analyzed (Participants) | 6270 | 6276
Percentage of participants
  MI | 1.52 | 1.78
  stroke | 1.20 | 1.07
  CV death* | 0.61 | 0.62
  UA | 0.32 | 0.32
  TIA | 0.67 | 0.72
Statistical Analysis 1: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of incidence of MI was conducted via a 2-sided log-rank test. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Other; p = 0.2325, Log Rank; Cox Proportional Hazard = 0.85, 95% CI 2-sided [0.64 to 1.11]
Statistical Analysis 2: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of incidence of stroke was conducted via a 2-sided log-rank test. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Other; p = 0.5072, Log Rank; Cox Proportional Hazard = 1.12, 95% CI [0.80 to 1.55]
Statistical Analysis 3: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of incidence of cardiovascular death was conducted via a 2-sided log-rank test. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Other; p = 0.9010, Log Rank; Cox Proportional Hazard = 0.97, 95% CI [0.62 to 1.52]
Statistical Analysis 4: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of incidence of UA was conducted via a 2-sided log-rank test. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Other; p = 0.9979, Log Rank; Cox Proportional Hazard = 1.00, 95% CI 2-sided [0.54 to 1.86]
Statistical Analysis 5: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of incidence of TIA was conducted via a 2-sided log-rank test. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Other; p = 0.7455, Log Rank; Cox Proportional Hazard = 0.93, 95% CI 2-sided [0.61 to 1.42]

7. Other Pre Specified Outcome: Number of Subjects With Adjudicated GI Bleeding by Severity
Time Frame: Until follow-up (approximate 6 years)
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) | Placebo
Number analyzed (Participants) | 6270 | 6276
Participants
  Total | 61 | 29
  Mild | 42 | 22
  Moderate | 15 | 5
  Severe | 4 | 2

8. Other Pre Specified Outcome: Incidence of Composite Outcomes and Non-fatal MI
Time Frame: Until follow-up (approximate 6 years)
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) | Placebo
Number analyzed (Participants) | 6270 | 6276
Percentage of participants
  MI, stroke, CV death, UA or TIA | 4.29 | 4.48
  MI, stroke or CV death | 3.32 | 3.47
  non-fatal MI | 1.40 | 1.56
Statistical Analysis 1: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of incidence of composite outcome of MI, stroke, CV death, UA or TIA was conducted via a 2-sided log-rank test. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Other; p = 0.6038, Log Rank; Cox Proportional Hazard = 0.96, 95% CI 2-sided [0.81 to 1.13]
Statistical Analysis 2: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of incidence of composite outcome of MI, stroke or CV death was conducted via a 2-sided log-rank test. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Other; p = 0.6190, Log Rank; Cox Proportional Hazard = 0.95, 95% CI 2-sided [0.79 to 1.15]
Statistical Analysis 3: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) vs Placebo; Analysis of incidence of non-fatal MI was conducted via a 2-sided log-rank test. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Other; p = 0.4562, Log Rank; Cox Proportional Hazard = 0.90, 95% CI 2-sided [0.67 to 1.20]

9. Other Pre Specified Outcome: Incidence of Composite Outcomes and Individual Outcomes in Per-protocol Population
Description: *all other CV death without fatal MI and fatal stroke.
Time Frame: Until follow-up (approximate 6 years)
Population: Per-protocol (PP) group (N=7702) consists of all patients who had no protocol violation.
Measure: Number; unit: Percentage of participants
Groups:
- Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol: Subjects received 1 tablet of enteric-coated acetylsalicylic acid [100 milligram (mg)] orally once daily.
- Placebo Per-protocol: Subjects received 1 tablets of matching placebo orally once daily.
Arm/Group | Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol | Placebo Per-protocol
Number analyzed (Participants) | 3790 | 3912
Percentage of participants
  MI, stroke, CV death, UA or TIA | 3.40 | 4.19
  MI, stroke or CV death | 2.72 | 3.45
  MI | 0.98 | 1.84
  Non-fatal MI | 0.84 | 1.53
  Stroke | 1.06 | 0.95
  CV death* | 0.69 | 0.66
  UA | 0.21 | 0.28
  TIA | 0.50 | 0.49
  All-cause mortality | 2.85 | 2.58
Statistical Analysis 1: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol vs Placebo Per-protocol; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.0756, Log Rank; Cox Proportional Hazard = 0.81, 95% CI 2-sided [0.64 to 1.02]
Statistical Analysis 2: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol vs Placebo Per-protocol; [analysis description as in outcome 8, analysis 2]; Test type: Other; p = 0.0661, Log Rank; Cox Proportional Hazard = 0.79, 95% CI 2-sided [0.61 to 1.02]
Statistical Analysis 3: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol vs Placebo Per-protocol; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.0014, Log Rank; Cox Proportional Hazard = 0.53, 95% CI 2-sided [0.36 to 0.79]
Statistical Analysis 4: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol vs Placebo Per-protocol; [analysis description as in outcome 8, analysis 3]; Test type: Other; p = 0.0056, Log Rank; Cox Proportional Hazard = 0.55, 95% CI 2-sided [0.36 to 0.84]
Statistical Analysis 5: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol vs Placebo Per-protocol; [analysis description as in outcome 6, analysis 2]; Test type: Other; p = 0.6291, Log Rank; Cox Proportional Hazard = 1.12, 95% CI [0.71 to 1.75]
Statistical Analysis 6: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol vs Placebo Per-protocol; Analysis of incidence of CV death was conducted via a 2-sided log-rank test. Results would be considered statistically significant if the 2-sided P value is ≤0.05; Test type: Other; p = 0.9161, Log Rank; Cox Proportional Hazard = 1.03, 95% CI 2-sided [0.60 to 1.77]
Statistical Analysis 7: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol vs Placebo Per-protocol; [analysis description as in outcome 6, analysis 4]; Test type: Other; p = 0.5380, Log Rank; Cox Proportional Hazard = 0.75, 95% CI [0.30 to 1.87]
Statistical Analysis 8: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol vs Placebo Per-protocol; [analysis description as in outcome 6, analysis 5]; Test type: Other; p = 0.9181, Log Rank; Cox Proportional Hazard = 1.03, 95% CI 2-sided [0.55 to 1.95]
Statistical Analysis 9: Comparison: Acetylsalicylic Acid (Aspirin, BAYE4465) Per-protocol vs Placebo Per-protocol; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.4796, Log Rank; Cox Proportional Hazard = 1.10, 95% CI 2-sided [0.84 to 1.45]

ADVERSE EVENTS:
Time Frame: Until follow-up (approximately 6 years)
Groups:
- Acetylsalicylic Acid: Subjects received 1 tablet of enteric-coated acetylsalicylic acid [100 milligram (mg)] orally one daily.
Arm/Group | Placebo | Acetylsalicylic Acid
Serious Adverse Events (participants affected / at risk) | 1311/6276 | 1266/6270
Other Adverse Events (participants affected / at risk) | 5053/6276 | 5059/6270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6276) | Acetylsalicylic Acid (N=6270)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 11 (11)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Accident at work (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 12 (12) | 10 (10)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (7) | 8 (8)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 58 (58) | 43 (44)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 2 (3)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (6)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Agitated depression (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 2 (2) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 2 (2)
Alcoholic liver disease (Hepatobiliary disorders) | 1 (1) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 3 (3)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (2)
Amaurosis fugax (Eye disorders) | 1 (1) | 2 (2)
Ameloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula infection (Infections and infestations) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 14 (15) | 20 (20)
Angina unstable (Cardiac disorders) | 19 (20) | 15 (17)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 9 (9) | 13 (13)
Aortic aneurysm (Vascular disorders) | 6 (6) | 10 (10)
Aortic aneurysm rupture (Vascular disorders) | 2 (2) | 2 (2)
Aortic dilatation (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 2 (2) | 0 (0)
Aortic stenosis (Vascular disorders) | 4 (4) | 0 (0)
Aortic valve calcification (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve disease mixed (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 4 (4) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 5 (5) | 3 (3)
Appendicitis (Infections and infestations) | 9 (10) | 9 (9)
Appendicitis perforated (Infections and infestations) | 3 (3) | 1 (1)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0)
Arteriogram coronary (Investigations) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (2) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (7)
Arthritis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 40 (41) | 37 (39)
Atrial flutter (Cardiac disorders) | 3 (3) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 4 (4) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 8 (8) | 0 (0)
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Axonal neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell unclassifiable lymphoma high grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 6 (6)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 2 (2)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Basilar artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 20 (20) | 10 (10)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 4 (4)
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary fistula (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biopsy prostate (Investigations) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 6 (6)
Bladder diverticulum (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder neck sclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Bladder sphincter atony (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (12) | 9 (10)
Bladder transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 2 (2)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 4 (4) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 2 (2) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 2 (2) | 2 (2)
Brain stem stroke (Nervous system disorders) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 10 (10)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 3 (3)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carcinoid tumour of the caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 9 (9) | 4 (4)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 7 (7)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 3 (3)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 9 (9) | 5 (5)
Carpal tunnel syndrome (Nervous system disorders) | 2 (3) | 1 (1)
Cataract (Eye disorders) | 5 (5) | 8 (10)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 8 (8) | 6 (6)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 3 (3) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral circulatory failure (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 3 (3)
Cerebral infarction (Nervous system disorders) | 5 (5) | 8 (9)
Cerebral ischaemia (Nervous system disorders) | 4 (4) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 9 (9) | 10 (10)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 2 (2)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chalazion (Eye disorders) | 1 (1) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest pain (General disorders) | 19 (19) | 23 (24)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 8 (9) | 13 (13)
Cholecystitis acute (Hepatobiliary disorders) | 8 (8) | 7 (7)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 17 (17) | 24 (24)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 4 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (11)
Chronic sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Circulatory collapse (Vascular disorders) | 3 (3) | 4 (4)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 14 (14)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Colon dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 2 (2)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Complex partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 6 (6)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital urinary tract obstruction (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Corneal degeneration (Eye disorders) | 0 (0) | 1 (1)
Corneal disorder (Eye disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 61 (63) | 46 (46)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (2)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 8 (8) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 2 (2) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dental operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 4 (6) | 3 (3)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 2 (2) | 1 (1)
Device loosening (Product Issues) | 4 (4) | 2 (2)
Device malfunction (Product Issues) | 0 (0) | 2 (2)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diffuse large B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 7 (8) | 5 (5)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 6 (6) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Dural abscess (Infections and infestations) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 6 (6)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Elbow operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Endocrine ophthalmopathy (Eye disorders) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 10 (11)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (2) | 2 (3)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extraskeletal myxoid chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eyelid dermatochalasis (Eye disorders) | 1 (1) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 2 (2)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 7 (8) | 4 (4)
Familial tremor (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 9 (10) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 3 (3) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (4)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fractured ischium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gallbladder enlargement (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gas poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 3 (3)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastroenteritis (Infections and infestations) | 4 (4) | 6 (6)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 13 (13)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal stromal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 2 (2)
Glaucoma (Eye disorders) | 3 (3) | 4 (4)
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 4 (4) | 6 (6)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 7 (7)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Haemophilia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 4 (4) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 4 (4)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Hemianaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (4) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Herpes zoster infection neurological (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster meningoencephalitis (Infections and infestations) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 4 (4) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 11 (12) | 2 (2)
Hydrocele (Congenital, familial and genetic disorders) | 2 (3) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 8 (8) | 3 (3)
Hypertensive crisis (Vascular disorders) | 11 (12) | 8 (10)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 2 (2) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incision site ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 4 (5) | 7 (11)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 31 (32) | 35 (35)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site injury (General disorders) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Insulinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (8)
Intestinal fibrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (4)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 2 (2) | 1 (1)
Intracranial haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 3 (3) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 19 (19) | 22 (22)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation reduction (Surgical and medical procedures) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Kidney contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 4 (4) | 0 (0)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Labile hypertension (Vascular disorders) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 3 (3) | 6 (6)
Lacunar stroke (Nervous system disorders) | 0 (0) | 2 (2)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 4 (6)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Laryngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (2)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukoplakia oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 4 (4)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (4)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (4) | 3 (3)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 10 (10)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 1 (1) | 1 (1)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 9 (9)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of pleura metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant nipple neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Medical device pain (General disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 2 (2) | 2 (2)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Meningitis meningococcal (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 11 (11) | 10 (10)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (2)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 4 (4) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0)
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Morton's neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Motor neurone disease (Nervous system disorders) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 2 (2)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Myocardial bridging (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 38 (38) | 29 (29)
Myocardial ischaemia (Cardiac disorders) | 10 (10) | 7 (7)
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 7 (7) | 6 (7)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgic amyotrophy (Nervous system disorders) | 1 (1) | 0 (0)
Neurodegenerative disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 2 (2)
Non-Hodgkin's lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Odontogenic cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Oral mucosal hypertrophy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 3 (3) | 0 (0)
Organ failure (General disorders) | 0 (0) | 1 (1)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 103 (109) | 104 (114)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (2) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Ovarian epithelial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Pancreas infection (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 5 (5)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 1 (1)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Parkinson's disease (Nervous system disorders) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Parotidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 2 (3) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Patient-device incompatibility (Product Issues) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (2)
Perihepatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 12 (12) | 5 (6)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 2 (2) | 1 (1)
Peripheral arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 3 (3) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 4 (4)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngeal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Phobia (Psychiatric disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleural calcification (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleuropericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 19 (19) | 26 (28)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Polyneuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Polypoidal choroidal vasculopathy (Eye disorders) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 2 (2)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 5 (5) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 44 (45) | 59 (59)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 5 (5)
Prostatic cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 2 (2)
Prostatism (Reproductive system and breast disorders) | 2 (3) | 4 (4)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 2 (2) | 4 (4)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 12 (12)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelocystitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Quadriparesis (Nervous system disorders) | 1 (1) | 0 (0)
Radicular syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 7 (7) | 2 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 6 (6)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Removal of internal fixation (Surgical and medical procedures) | 2 (2) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Renal colic (Renal and urinary disorders) | 8 (8) | 8 (8)
Renal cyst (Renal and urinary disorders) | 2 (2) | 1 (4)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Retinal artery embolism (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 2 (2) | 0 (0)
Retinal detachment (Eye disorders) | 3 (4) | 3 (3)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinophyma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 13 (13) | 6 (6)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 3 (3) | 2 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (2) | 1 (1)
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 6 (6) | 4 (5)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Serum ferritin increased (Investigations) | 1 (1) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (2)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal vascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (2)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Strabismus (Eye disorders) | 1 (1) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (2)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (2)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 3 (3)
Sudden cardiac death (General disorders) | 1 (1) | 2 (2)
Sudden death (General disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 2 (2)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 12 (13) | 7 (7)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 2 (2)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Testicular disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testis discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (2) | 1 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosed varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Thyroid cyst (Endocrine disorders) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 3 (3)
Transient global amnesia (Nervous system disorders) | 3 (3) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 30 (31) | 26 (27)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Tympanoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 (7) | 8 (8)
Type IIa hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 4 (4) | 5 (5)
Unevaluable event (General disorders) | 1 (1) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary bladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 8 (8) | 6 (7)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 9 (9)
Urine flow decreased (Renal and urinary disorders) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 4 (4) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Uterovaginal prolapse (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Uveitis-glaucoma-hyphaema syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VIIIth nerve lesion (Nervous system disorders) | 1 (1) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
VIth nerve paresis (Nervous system disorders) | 1 (1) | 0 (0)
Vaginal haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 5 (5)
Vaginal prolapse repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 8 (9) | 5 (5)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 4 (4) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 3 (3) | 1 (1)
Wernicke's encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Yersinia infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6276) | Acetylsalicylic Acid (N=6270)
Arthralgia (Musculoskeletal and connective tissue disorders) | 653 (803) | 636 (816)
Back pain (Musculoskeletal and connective tissue disorders) | 688 (908) | 695 (897)
Bronchitis (Infections and infestations) | 482 (680) | 514 (741)
Cough (Respiratory, thoracic and mediastinal disorders) | 497 (601) | 442 (556)
Dyspepsia (Gastrointestinal disorders) | 362 (419) | 374 (446)
Hypertension (Vascular disorders) | 514 (578) | 478 (526)
Lower respiratory tract infection (Infections and infestations) | 420 (703) | 377 (650)
Nasopharyngitis (Infections and infestations) | 407 (524) | 421 (550)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 423 (517) | 468 (548)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 359 (406) | 354 (406)
Upper respiratory tract infection (Infections and infestations) | 371 (491) | 348 (443)
Urinary tract infection (Infections and infestations) | 321 (474) | 363 (549)

LIMITATIONS AND CAVEATS:
The reported analyses are limited to endpoint events that met strict criteria. Further blinded review of events is ongoing to identify endpoints based on pragmatic criteria. Interpretations for clinical decision making should await future reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days